CLINICAL TRIAL: NCT06481345
Title: Characterization of Myeloproliferative Neoplasia With a Mutated IDH, SRSF2 or SF3B1 Allele
Brief Title: Characterization of Myeloproliferative Neoplasia With a Mutated IDH, SRSF2 or SF3B1 Allele (CARPEDIEM)
Acronym: CARPEDIEM
Status: Active, not recruiting | Type: Observational
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: 29BRC24.0154 - CARPEDIEM
Record Dates: First submitted 2024-06-25; First posted 2024-07-01 (Actual); Last update posted 2024-07-01 (Actual); Status verified 2024-04

CONDITIONS: Myeloproliferative Disorders
MeSH Terms: conditions — Myeloproliferative Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- MPN patients with IDH1/2 mutation
- MPN patients with SRSF2 mutation
- MPN patients with SF3B1 mutation

SUMMARY:
Retrospective study assessing the impact of IDH1/2, SRSF2 or SF3B1 mutations on event free survival of MPN patients

DETAILED DESCRIPTION:
Patients with a diagnosis of MPN and a mutation of IDH1/2, SRSF2 or SF3B1 will be included. Clinical and biological characterisation at diagnosis, as well as evlution will be recorded. Event free survival will be assessed in each group (event = thrombosis, transformation to mylofibrosis/acute leukemia, death).

ELIGIBILITY:
Inclusion Criteria:

* Patients with MPN diagnosis
* Mutation in IDH1/2, SRSF2 or SF3B1

Exclusion Criteria:

* Unable to consent

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients followed by hematologists of the French Intergroup of MPN
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2024-06-25 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Event free survival | 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Brest, Brest, France

IPD SHARING:
Plan to Share IPD: Yes
All collected data that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: Data will be available beginning three years and ending fifteen years following the final study report completion
Access Criteria: Data access requests will be reviewed by the internal committee of Brest UH. Requestors will be required to sign and complete a data access agreement